CLINICAL TRIAL: NCT01565369
Title: Evaluation of Physician Training for Interpretation of Florbetapir-PET Scans: Validation of Binary Image Rating Methodology Using Amyloid Histopathology at Autopsy as the Reference Standard.
Brief Title: Evaluation of Physician Training Methods to Read Florbetapir-PET Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A08
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
The purpose of this study is re-read of brain amyloid positron emission tomography (PET) scans acquired in previous florbetapir F 18 clinical studies by readers trained using updated reading methodology. The scans in this study came from subjects who had an autopsy to reveal the subject's true amyloid status.

ELIGIBILITY:
Inclusion Criteria (Study A07[NCT00857415]):

* Have a projected life expectancy of ≤ 6 months as determined by the principal investigator (e.g. terminal medical condition) or are already enrolled in a longitudinal study of aging with an autopsy component;
* Can tolerate a 10 minute PET scan; and
* Give informed consent for study procedures and brain donation consistent with the legal requirements of the State in which they are enrolled and the State in which they die.

Exclusion Criteria (Study A07[NCT00857415]):

* Have primary brain tumor, known metastases to the brain, central nervous system (CNS) lymphoma;
* Have any major, focal structural loss of brain matter;
* Are aggressively being treated with life sustaining measures (e.g. currently on respirator; receiving high dose chemotherapy);
* Have a clinically significant infectious disease, including Acquired Immune Deficiency Syndrome (AIDS), Human Immunodeficiency Virus (HIV) infection, previous positive test for hepatitis or HIV or Creutzfeldt-Jakob disease (CJD);
* Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
* Have ever participated in an experimental study with an amyloid targeting agent (e.g. anti-amyloid immunotherapy, secretase inhibitor);
* Have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session; or
* Are females of childbearing potential who are pregnant or not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NO SUBJECTS WERE ENROLLED IN THIS STUDY - this study re-read scans obtained in other clinical studies
Groups:
- All A07 Autopsy Subjects: Subjects who had a valid florbetapir-PET scan and came to autopsy in Study A07
Period: Overall Study
Arm/Group | All A07 Autopsy Subjects
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All A07 Autopsy Subjects
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 79.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Florbetapir PET Scans to Detect Moderate to Frequent Amyloid Plaque
Description: Nine readers blinded to all clinical information using the binary read methodology (amyloid positive/negative). Sensitivity will be calculated as the percent of true positives (as determined by the reference standard, moderate or frequent amyloid plaque at autopsy) that are correctly identified as amyloid positive by the PET scan read. Reported as the median sensitivity of the nine readers.
Time Frame: 50-60 min after injection
Population: 19 of the 35 subjects had moderate or frequent plaques at autopsy
Measure: Median (Full Range); unit: percentage of true positives
Groups:
- All A07(NCT00857415) Autopsy Subjects: Subjects who had a valid florbetapir-PET scan and came to autopsy in Study A07(NCT00857415)
Arm/Group | All A07(NCT00857415) Autopsy Subjects
Number analyzed (Participants) | 19
percentage of true positives | 100 [84.2 to 100]

2. Primary Outcome: Specificity of Florbetapir PET Scans to Detect Moderate to Frequent Amyloid Plaque
Description: Nine readers blinded to all clinical information using the binary read methodology (amyloid positive/negative). Specificity will be calculated as the percent of true negatives (as determined by the reference standard, no or sparse amyloid plaque at autopsy) that are correctly identified as amyloid negative by the PET scan read. Reported as the median specificity of the nine readers.
Time Frame: 50-60 min after injection
Population: 16 of the 35 subjects had none or sparse plaques at autopsy
Measure: Median (Full Range); unit: percentage of true negatives
Groups:
- All A07 Autopsy Subjects: Subjects who had a valid florbetapir-PET scan and came to autopsy in Study A07(NCT00857415)
Arm/Group | All A07 Autopsy Subjects
Number analyzed (Participants) | 16
percentage of true negatives | 93.8 [68.8 to 100]

3. Secondary Outcome: Inter-reader Agreement
Description: Percentage of individual scan reads that agreed or disagreed with the majority read across nine readers
Time Frame: 50-60 min after injection
Population: 315 scans = 35 subjects x 9 readers
Measure: Number; unit: percentage of scans
Units Other Than Participants: florbetapir PET scan reads
Arm/Group | All A07(NCT00857415) Autopsy Subjects
Number analyzed (Participants) | 35
Number analyzed (florbetapir PET scan reads) | 315
percentage of scans
  Agreed with majority read | 96.2
  Discrepant with majority read | 3.8
Statistical Analysis 1: Comparison: All A07(NCT00857415) Autopsy Subjects; Fleiss' kappa; Test type: Superiority or Other; p < 0.0001, Fleiss' kappa — evaluated at the .05 significance level; Fleiss' kappa = 0.8547, Standard Error of Mean 0.0282

ADVERSE EVENTS:
Description: No subjects received florbetapir in this study. This study consisted of rereads of scans previously acquired in another clinical study (A07).
Arm/Group | All A07 Autopsy Subjects
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days